CLINICAL TRIAL: NCT05186311
Title: A Prospective Multi-center Study to Evaluate Clinical Equivalence (Method Comparison) Between the BD MiniDraw™ SST™ Capillary Blood Collection Tube and BD MiniDraw™ EDTA Capillary Blood Collection Tube to Respective Comparators
Brief Title: BD MiniDraw™ Capillary System Clinical Equivalence Study
Status: Completed | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: Babson Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAS-21YODA005
Record Dates: First submitted 2021-12-17; First posted 2022-01-11 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Healthy; Disease, Chronic; Acute Disease; Sample Collection
Keywords: sample collection device
MeSH Terms: conditions — Chronic Disease; Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Test product (Experimental): BD MiniDraw™ Capillary Blood Collection System
  Interventions: Device: Capillary Blood Collection System

INTERVENTIONS:
Device: Capillary Blood Collection System — Test Blood Sample Collection
  Other Names: BD MiniDraw™ Capillary System

SUMMARY:
This study designed to evaluate the safety and effectiveness of a newly developed sample collection device. Participants will be enrolled and samples will be collected by representative future users of the device. Comparator venous and conventional capillary tubes will be collected by skilled healthcare professionals with phlebotomy experience. Samples will be tested and average differences between the investigational device compared to a marketed comparator will be evaluated. Visual observations will be captured and device safety will be assessed.

DETAILED DESCRIPTION:
The current method for collection of a large volume of capillary blood (up to 600 µL) involves optional warming of the hand or finger prior to procedure, lancing of the fingertip, squeezing the fingertip by hand, and dripping the blood into an open non-sterile tube. The capillary blood collection process is considered cumbersome and lacks standardization in how much pressure is applied in squeezing of the finger which may lead to poor sample quality or insufficient blood volume. Common sample quality issues for capillary blood collection include hemolysis and dilution of sample with interstitial fluid, potentially causing bias in test results. Open collection also carries a risk of blood exposure for healthcare workers and potential risk of infection at the finger puncture site. A new device, BD Microtainer® Easy Collect Capillary Blood Collection System for the collection of capillary blood was created to standardize the current collection process and improve sample quality.

This study designed to evaluate the safety and effectiveness of the BD Microtainer® Easy Collect Capillary Tube SST™ and BD Microtainer® Easy Collect Capillary Tube EDTA devices. This study will be conducted in two parts, one for the SST product and the other for the EDTA product. A minimum of 100 participants, and a maximum of 150 participants per part will be enrolled at a minimum of three various ancillary healthcare site settings representative of the intended use environment such as retail pharmacy site, patient service center, and/or urgent care clinic. Samples will be collected by representative future users of the BD Microtainer® Easy Collect Capillary Blood Collection System who may not have prior blood collection experience. Comparator venous and conventional capillary tubes will be collected by skilled healthcare professionals with phlebotomy experience. Samples will be collected, clotted (serum samples only) and centrifuged (serum samples only) before transportation to the laboratory where they will be tested.

Average differences between the investigational device compared to a marketed comparator will be evaluated. Visual observations for the SST products will be captured which include hemolysis as measured by Plasma Free Hemoglobin (PFH); collection volume; and duration of sample collection. Visual Observations for the EDTA products will be captured which include frequency of occurrence of instrument flags; frequency of occurrence of platelet clump instrument flags; frequency of instrument platelet clump flags with no platelet clump; evaluate whole blood collection volume; and duration of sample collection. Lastly, device safety will be assessed by device and procedure related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age.
* Not currently pregnant (self-reported)
* Adequate access to four fingers (ring and middle finger on each hand) and inner elbows for blood collection procedures
* Willing and able to comply with all study procedures and evaluations
* Ability to read, write, and understand English language
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Evidence of skin issues such as infections, ulcerations, blisters, peripheral vascular disease, inflammation, extensive scarring or calluses, or healed burns at the fingerstick site. Subject to post-study exclusion period for this or other related studies:

  1. A study participant may enroll once in study part A and once in study part B of this clinical study. They may not enroll more than once in a single study part.
  2. If a study participant has previously enrolled in one study part and would like to enroll in the second study part, they must wait 8 days from the time of the first study part collection procedures to enroll in the second study part collection procedures.
* Any condition which, in the opinion of the Investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Babson Diagnostics, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Part A: Serum
Arm/Group | Test Product
Started | 136
Completed | 135
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Part B: EDTA
Arm/Group | Test Product
Started | 126
Completed | 125
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Test Product
Number analyzed (Participants) | 262
Age, Customized [Count of Participants; unit: Participants]
  Age over 18 | 262
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 149
  Sex/Gender: Male | 96
  Sex/Gender: not reported | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Chemistry Analytes [Albumin (ALB) and Total Protein (TP)] in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of g/dL
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: g/dL
Units Other Than Participants: Blood Sample
Arm/Group | Test Product
Number analyzed (Participants) | 100
Number analyzed (Blood Sample) | 102
g/dL
  ALB Test Device SST™ | 3.746 [1.01 to 5.54]
  ALB Capillary Comparator SST™ | 3.787 [1.01 to 5.58]
  TP Test Device SST™ | 6.77 [2.6 to 10.2]
  TP Capillary Comparator SST™ | 6.83 [2.7 to 10.2]
  ALB Venous comparator Serum | 3.791 [1.00 to 5.44]
  TP Venous comparator Serum | 6.78 [2.6 to 9.8]
Statistical Analysis 1: Comparison: Test Product; One hundred (100) participants (with paired numerical data) per each analyte provide > 90% power to ensure that mean biases and confidence intervals are within the clinical acceptance limit (CAL), at medically relevant points, assuming no true bias between the tube types, residual standard deviation (SD) or coefficient of variation (CV) = CAL and collected data cover medically relevant points; Test type: Equivalence — The estimated regression equation was then used to estimate the bias (with two one-sided 95% confidence intervals, referred to as 95% limits in the text) between the evaluation tube and the comparator tube at all prespecified medical decision levels. The biases and 95% limit were compared to the clinical acceptance limit (CAL); No p-value were established. Rather a bias between tube types at pre-determined medical decision points were estimated with 95% intervals. The mean biases and 95% limit were compared to the CAL. For equivalence testing the initial alpha level is set at 10%. This corresponds to obtaining 90% confidence intervals (associated with 95% two 1-sided confidence limits). Since the clinical equivalence includes two comparisons, the actual alpha used for each comparison was set to 5%, using a Bonferroni correction. No other adjustment for multiplicity will be made on any other comparisons. Note that for the confidence intervals (CI) calculated for the intercept and slope of the regression parameters, no multiplicity adjustments on the a level are performed (alpha = 0.05)

2. Primary Outcome: White Blood Cell Differential Counts, Hemoglobin A1c, Hematocrit, and Red Blood Cell Distribution Width in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators venous comparator and capillary comparator. This comparison was focused on the analytes with a unit of percentage
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: % of analyte in the sample
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 117
% of analyte in the sample
  Basophils (BA)% Test Device EDTA | 0.73 [0.0 to 2.0]
  BA% Capillary Comparator EDTA | 0.71 [0.0 to 1.9]
  BA% Venous comparator EDTA | 0.71 [0.0 to 1.8]
  Eosinophils (EO)% Capillary Comparator EDTA | 2.97 [0.0 to 12.0]
  EO% Venous comparator EDTA | 3.16 [0.0 to 16.0]
  EO% Test Device EDTA | 2.89 [0.0 to 10.7]
  hemoglobin A1c (HbA1c) Capillary Comparator EDTA | 5.938 [4.20 to 14.20]
  HbA1c Venous comparator EDTA | 5.965 [4.60 to 14.10]
  HbA1c Test Device EDTA | 5.934 [4.20 to 14.20]
  HCT Capillary Comparator EDTA | 39.41 [19.2 to 73.6]
  Hematocrit (HCT) Venous comparator EDTA | 39.26 [18.5 to 73.8]
  HCT Test Device EDTA | 39.9 [19.1 to 73.1]
  Lymphocytes (LY)% Capillary Comparator EDTA | 27.93 [7.2 to 67.7]
  LY% Venous comparator EDTA | 27.85 [7.4 to 67.2]
  LY% Test Device EDTA | 27.69 [6.8 to 67.5]
  Monocytes (MO)% Capillary Comparator EDTA | 8.4 [3.8 to 22.3]
  MO% Venous comparator EDTA | 8.49 [4.0 to 19.4]
  MO% Test Device EDTA | 8.6 [4.2 to 20.7]
  Neutrophils (NE)% Capillary Comparator EDTA | 59.51 [9.5 to 84.3]
  NE% Venous comparator EDTA | 59.39 [9.2 to 84.4]
  NE% Test Device EDTA | 59.7 [10.5 to 84.2]
  Red Blood Cell Distribution Width (RDW)-CV Capillary Comparator EDTA | 13.54 [11.4 to 24.0]
  RDW-CV Venous comparator EDTA | 13.67 [11.4 to 23.9]
  RDW-CV Test Device EDTA | 13.55 [11.4 to 24.0]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — The estimated regression equation was then used to estimate the bias (with two one-sided 95% confidence intervals, referred to as 95% limits in the text) between the evaluation tube and the comparator tube at all prespecified medical decision levels. The biases and 95% limit were compared to the clinical acceptance limit; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Thyroid Stimulating Hormone (TSH) in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of µIU/mL
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: µIU/mL
Arm/Group | Test Product
Number analyzed (Participants) | 94
µIU/mL
  TSH Test Device SST™ | 4.7599 [0.183 to 97.892]
  TSH Capillary Comparator SST™ | 5.4529 [0.181 to 104.351]
  TSH Venous comparator Serum | 5.4211 [0.188 to 101.313]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Lipid Analytes and Metabolic Analytes, in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of mg/dL
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Test Product
Number analyzed (Participants) | 102
mg/dL
  blood urea nitrogen (BUN) Test Device SST™ | 21.9 [8 to 115]
  BUN Capillary Comparator SST™ | 22 [7 to 115]
  Calcium (Ca) Test Device SST™ | 9.43 [2.7 to 13.6]
  Ca Capillary Comparator SST™ | 9.52 [2.7 to 13.5]
  cholesterol (Chol) Test Device SST™ | 190.2 [51 to 454]
  Chol Capillary Comparator SST™ | 192.8 [51 to 457]
  Creatinine (Creat) Test Device SST™ | 2.418 [0.23 to 19.93]
  Creat Capillary Comparator SST™ | 2.432 [0.22 to 20.03]
  Glucose (GLUC) Test Device SST™ | 158.2 [36 to 1434]
  GLUC Capillary Comparator SST™ | 159.1 [37 to 1443]
  high-density lipoprotein (HDL) Test Device SST™ | 51.28 [21.5 to 96.0]
  HDL Capillary Comparator SST™ | 52.54 [21.7 to 99.5]
  low-density lipoprotein (LDL) Test Device SST™ | 131.07 [32.8 to 612.4]
  LDL Capillary Comparator SST™ | 132.76 [33.1 to 609.2]
  Total Bilirubin (TBIL) Test Device SST™ | 1.8604 [0.170 to 26.420]
  TBIL Capillary Comparator SST™ | 1.8763 [0.180 to 26.519]
  Triglycerides (Trig) Test Device SST™ | 155 [32 to 730]
  Trig Capillary Comparator SST™ | 158.6 [33 to 739]
  BUN Venous comparator Serum | 20.4 [6 to 115]
  Ca Venous comparator Serum | 9.51 [2.9 to 13.6]
  Chol Venous comparator Serum | 195.8 [59 to 456]
  Creat Venous comparator Serum | 2.11 [0.22 to 19.87]
  GLUC Venous comparator Serum | 149.4 [36 to 1428]
  HDL Venous comparator Serum | 54.83 [21.5 to 109.6]
  LDL Venous comparator Serum | 140.78 [35.1 to 610.6]
  TBIL Venous comparator Serum | 1.7931 [0.180 to 26.653]
  Trig Venous comparator Serum | 157.9 [32 to 739]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

5. Primary Outcome: Metabolic Analytes, in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of mmol/L
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: mmol/L
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 102
Number analyzed (Blood samples) | 102
mmol/L
  chloride (CL) Test Device SST™ | 107.37 [73.2 to 146.0]
  CL Capillary Comparator SST™ | 107.11 [73.0 to 145.0]
  Carbon Dioxide (CO2) Test Device SST™ | 21.72 [14.0 to 33.8]
  CO2 Capillary Comparator SST™ | 24.02 [16.0 to 34.2]
  potassium (K) Test Device SST™ | 4.436 [2.14 to 8.15]
  K Capillary Comparator SST™ | 4.506 [2.12 to 8.10]
  Sodium (Na) Test Device SST™ | 138.29 [90.8 to 166.0]
  Na Capillary Comparator SST™ | 139.08 [90.9 to 166.0]
  CL Venous comparator Serum | 104.94 [72.4 to 145.0]
  CO2 Venous comparator Serum | 28.2 [16.4 to 35.2]
  K Venous comparator Serum | 4.228 [2.15 to 8.16]
  Na Venous comparator Serum | 139.33 [92.4 to 166.0]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

6. Primary Outcome: Vitamin D (Vit D), in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of ng/mL
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: ng/mL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 99
Number analyzed (Blood samples) | 99
ng/mL
  Vit D Test Device SST™ | 41.784 [10.11 to 103.56]
  Vit D Capillary Comparator SST™ | 36.786 [8.33 to 90.78]
  Vit D Venous comparator Serum | 37.603 [8.31 to 99.74]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

7. Primary Outcome: Alkaline Phosphatase (ALP), Alanine Transaminase (ALT), and Aspartate Aminotransferase (AST), in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To demonstrate clinical equivalence of the SST test device as compared to Venous Comparator Serum and Capillary Comparator for chemistry analytes. This comparison was focused on the analytes with a unit of U/L
Time Frame: within 4 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: U/L
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 97
Number analyzed (Blood samples) | 97
U/L
  ALKP Test Device SST™ SST™ | 98.6 [31 to 644]
  ALKP Capillary Comparator SST™ | 98.9 [31 to 646]
  ALT Test Device SST™ | 50.2 [8 to 756]
  ALT Capillary Comparator SST™ | 51 [8 to 759]
  AST Test Device SST™ | 47.4 [11 to 717]
  AST Capillary Comparator SST™ | 49.5 [10 to 719]
  ALKP Venous comparator Serum | 100.4 [31 to 649]
  ALT Venous comparator Serum | 50.4 [9 to 760]
  AST Venous comparator Serum | 45.7 [10 to 720]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

8. Primary Outcome: White Blood Cells (WBC) and Platelets (PLT) in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators Venous Comparator and Capillary Comparator. This comparison was focused on the analytes with a unit of 10^3/µL
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: 10^3 cells per µL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 117
10^3 cells per µL
  PLT Capillary Comparator EDTA | 275.3 [33 to 2967]
  PLT Venous comparator EDTA | 297 [34 to 2978]
  PLT Test Device EDTA | 262.1 [31 to 2964]
  WBC Capillary Comparator EDTA | 12.647 [2.28 to 267.31]
  WBC Venous comparator EDTA | 12.453 [2.01 to 265.52]
  WBC Test Device EDTA | 12.746 [2.39 to 265.50]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

9. Primary Outcome: Red Blood Cells (RBC) in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators Venous Comparator and Capillary Comparator. This comparison was focused on the analytes with a unit of 10^6/µL
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: 10^6 cells per µL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 117
10^6 cells per µL
  RBC Capillary Comparator EDTA | 4.43 [1.93 to 8.60]
  RBC Venous comparator EDTA | 4.375 [1.87 to 8.62]
  RBC Test Device EDTA | 4.471 [1.93 to 8.50]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

10. Primary Outcome: Mean Corpuscular Volume (MCV) and Red Blood Cell Distribution Width (RDW) in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators Venous Comparator and Capillary Comparator. This comparison was focused on the analytes with a unit of fL
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: fL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 108
fL
  MCV Capillary Comparator EDTA | 89.38 [75.9 to 104.4]
  MCV Venous comparator EDTA | 90.16 [75.5 to 104.4]
  MCV Test Device EDTA | 89.66 [75.6 to 104.6]
  RDW-SD Capillary Comparator EDTA | 44.14 [36.3 to 86.9]
  RDW-SD Venous comparator EDTA | 44.97 [37.3 to 86.0]
  RDW-SD Test Device EDTA | 44.32 [36.5 to 84.5]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

11. Primary Outcome: Hemoglobin (HgB) and Mean Corpuscular Hemoglobin Concentration (MCHC) in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators Venous Comparator and Capillary Comparator. This comparison was focused on the analytes with a unit of g/dL
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: g/dL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 117
g/dL
  HGB Capillary Comparator EDTA | 13.33 [6.2 to 25.5]
  HGB Venous comparator EDTA | 13.13 [6.1 to 25.4]
  HGB Test Device EDTA | 13.45 [6.2 to 25.3]
  MCHC Capillary Comparator EDTA | 33.81 [31.2 to 36.6]
  MCHC Venous comparator EDTA | 33.4 [30.7 to 36.2]
  MCHC Test Device EDTA | 33.69 [31.5 to 36.3]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

12. Primary Outcome: Mean Corpuscular Hemoglobin (MCH) in Plasma Measured With Ethylenediaminetetraacetic Acid (EDTA)
Description: To demonstrate clinical equivalence of the EDTA test device as compared to their relevant comparators Venous Comparator and Capillary Comparator. This comparison was focused on the analytes with a unit of pg
Time Frame: within 2 hours of sample collection
Population: This was a test for an analyte result. If there was no measurable value reported, it was not included in the analysis.
Measure: Mean (Full Range); unit: pg
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 126
Number analyzed (Blood samples) | 108
pg
  MCH Capillary Comparator EDTA | 30.22 [24.1 to 36.6]
  MCH Venous comparator EDTA | 30.12 [23.5 to 36.4]
  MCH Test Device EDTA | 30.21 [24.4 to 35.9]
Statistical Analysis 1: Comparison: Test Product; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; [other analysis details as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Plasma Free Hemoglobin (PFH) in Serum Measured Using the Silica Clot Activator for Serum Samples
Description: To evaluate sample hemolysis as measured by Plasma Free Hemoglobin (PFH) for BD Microtainer® Easy Collect Capillary Tube SST™ and all comparator tube types: capillary and venous
Time Frame: within 4 hours of sample collection
Measure: Mean (95% Confidence Interval); unit: mg/dL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 135
Number analyzed (Blood samples) | 254
mg/dL
  Test Device SST™ | 20.2659 [18.1190 to 22.4129]
  Capillary Comparator SST™ | 44.9719 [38.9098 to 51.0339]
  Venous comparator SST™ | 11.2487 [10.0577 to 12.4397]
  Venous comparator Serum | 9.8032 [8.3323 to 11.2742]

14. Other Pre Specified Outcome: Serum Collection Volume of the Test Device SST Tube
Description: To evaluate serum collection volume of the Test Device SST tube
Time Frame: within 4 hours of sample collection
Population: samples for collection volume
Measure: Mean (95% Confidence Interval); unit: uL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 135
Number analyzed (Blood samples) | 208
uL | 236.41521 [231.51278 to 241.31763]

15. Other Pre Specified Outcome: Duration of Sample Collection for Test Device SST Tube and Comparator Tube
Description: To evaluate duration of sample collection for Test Device SST tube tube and capillary comparator.
Time Frame: within 4 hours of sample collection
Population: time to fill tube
Measure: Mean (95% Confidence Interval); unit: seconds
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 135
Number analyzed (Blood samples) | 222
seconds
  Capillary Comparator SST™ | 108.7 [99.3 to 118.1]
  Test Device SST™ | 128.0 [117.5 to 138.6]

16. Other Pre Specified Outcome: Frequency of Occurrence of All Instrument Flags (Both Asterisks and IP Messages) in the Test Device EDTA and All Comparator Tube Types
Description: Evaluation of the frequency of occurrence of all instrument flags (both asterisks and IP messages) in the Test Device EDTA and all comparator tube types: venous and capillary tubes
Time Frame: within 4 hours of sample collection
Population: samples from tubes collected from participants.
Measure: Count of Units; unit: Blood samples
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 135
Number analyzed (Blood samples) | 124
Blood samples
  Test Device EDTA | 30
  Capillary Comparator EDTA: number analyzed (Blood samples) | 118
  Capillary Comparator EDTA | 25
  BD Venous comparator EDTA: number analyzed (Blood samples) | 122
  BD Venous comparator EDTA | 5
  Venous comparator EDTA: number analyzed (Blood samples) | 121
  Venous comparator EDTA | 5

17. Other Pre Specified Outcome: Whole Blood Collection Volume for the Test Device EDTA
Description: To evaluate whole blood collection volume for the Test Device EDTA
Time Frame: within 4 hours of sample collection
Population: samples from tubes collected
Measure: Mean (95% Confidence Interval); unit: uL
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 125
Number analyzed (Blood samples) | 121
uL | 299.37786 [290.6445 to 308.11119]

18. Other Pre Specified Outcome: Duration of Sample Collection for the Test Device EDTA and Capillary Comparator
Description: To evaluate duration of sample collection for the Test Device EDTA and capillary comparator
Time Frame: within 4 hours of sample collection
Population: samples from tubes filled
Measure: Mean (Full Range); unit: s
Units Other Than Participants: Blood samples
Arm/Group | Test Product
Number analyzed (Participants) | 125
Number analyzed (Blood samples) | 121
s
  Capillary Comparator EDTA | 95.8 [84.7 to 106.8]
  Test Device EDTA | 81 [72.8 to 89.2]

ADVERSE EVENTS:
Time Frame: 7 days
Description: Adverse events did not differ from the Clinicaltrials.gov definitions. A minimal number of adverse events, if any, would was expected for this study.
Groups:
- Comparator Product: respective comparator
  Comparator Blood Collection system: Comparator Blood Collection system
Arm/Group | Test Product | Comparator Product
All-Cause Mortality (participants affected / at risk) | 0/262 | 0/262
Serious Adverse Events (participants affected / at risk) | 0/262 | 0/262
Other Adverse Events (participants affected / at risk) | 0/262 | 0/262

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05186311/Prot_SAP_003.pdf